CLINICAL TRIAL: NCT05371808
Title: An Economic Analysis of Early vs Delayed Therapy in Newly Diagnosed Asymptomatic High-Risk Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma: A Companion Analysis to CCTG CLC.3/SWOG 1925 Randomized Phase III Clinical Trial
Brief Title: Economic Analysis of Early vs Delayed Therapy in Newly Diagnosed Asymptomatic High-Risk Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma:
Status: Recruiting | Type: Observational
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CLC3E
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: EQ-5D-5L Instrument — This instrument is a measure of health status for use in evaluating health and healthcare.
Other: Work Productivity and Daily Activity Impairment (WPAI) survey — The questionnaire includes three open-ended questions that determines: 1) hours absent from work due to health problems; 2) hours absent from work due to other reasons; and (3) hours actually worked over the past 30 days. Additional questions ask about the impact of health problems on work productivity and daily activities and are scored along a vertical visual analog scale. The WPAI provides estimates on absenteeism, presenteeism, global measures of lost productivity (absenteeism+presenteeism) and daily activity impairment (impaired ability to perform non-work activities including work around the house, child care, exercise, studying, and leisure activities)
Other: Resource Utilization Form (SMRC) — Resource utilization data collection will be supplemented by a self-administered resource utilization form (Stanford SMRC) to document non-protocol specified utilization. This will include hospitalizations (including days in hospital), emergency room visits, and non-protocol specified ambulatory visits.

SUMMARY:
Utilization data will be collected from all patients entered on the trial at Canadian centres from the time of registration until death, removal from study, or completion of 10 years of follow-up.

Protocol-specified health care utilization will be collected within trial case report forms, and will include study visits, radiographic assessments, laboratory investigations, and treatment administration.

Resource utilization data collection will be supplemented by a self-administered resource utilization form (Stanford SMRC) to document non-protocol specified utilization. This will include hospitalizations (including days in hospital), emergency room visits, and non-protocol specified ambulatory visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be eligible for the core CLC3/S1925 protocol.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life and/or health utility questionnaires in either English or French. The baseline assessment must be completed within required timelines, prior to enrollment. Inability (lack of comprehension in English or French, or other equivalent reason such as cognitive issues or lack of competency) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible.
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Canadian patients who are eligible for the core protocol CLC3/S1925 will be mandated to participate in the companion study CLC.3E.
  This study is designed to include women and minorities as appropriate, but is not designed to measure differences in intervention effects.
Sampling Method: Probability Sample
Enrollment: 247 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
To determine incremental cost-utility ratio of an early novel therapy approach compared to a deferred approach in Canadian patients with high-risk CLL (enrolled in the randomized component of the SWOG S1925/CLC3 study). | 10 years
  Direct medical costs will be estimated from the perspective of the Canadian public healthcare system. The denominator of the ratio will be expressed in quality-adjusted life years gained.

SECONDARY OUTCOMES:
To determine incremental cost-effectiveness ratio of an early novel therapy approach compared to a deferred approach in Canadian patients with high-risk CLL . Effectiveness will be expressed in life years gained | 10 years
To determine the incremental cost-effectiveness ratio of an early novel therapy approach compared to a deferred approach in Canadian patients with high-risk CLL. Effectiveness will be expressed in years prior to second progression gained. | 10 years
To determine the direct medical costs associated with the care of Canadian high-risk CLL patients randomized to an early treatment approach compared to a deferred approach. | 10 years
To compare the change in health preference (utility) over time for individuals with high-risk CLL randomized to an early approach vs. deferred treatment approach | 10 years
To compare the lost productivity for Canadian individuals with high-risk CLL randomized to an early treatment approach compared to a deferred approach | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cheung, Study Chair — Odette Cancer Centre, Sunnybrook Helath Sciences Centre, Toronto, Ontario, Canada
Locations (8):
- Canada (8):
  - BCCA - Vancouver, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - The Jewish General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No